CLINICAL TRIAL: NCT05036174
Title: Diphenhydramine 5% Ointment for Pain in Knee Osteoarthritis: a Randomised Double-blind Placebo-controlled Pilot Feasibility Study
Brief Title: Diphenhydramine Ointment for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology (Other)
Responsible Party: Principal Investigator, Ivan Shirinsky, MD, PhD, Head of the laboratory of immunopharmacology, Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 415-5.13.04.2021-1
Record Dates: First submitted 2021-06-08; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; pain; antihistamines
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diphenhydramine (Experimental): Topical 5% diphenhydramine ointment applied at knee joint at a dose of 2 g three times a day for 7 days
  Interventions: Drug: Diphenhydramine 5%
- Placebo (Placebo Comparator): Vehicle (placebo) ointment applied at knee joint at a dose of 2 g three times a day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diphenhydramine 5% — Diphenhydramine 5% ointment
  Arms: Diphenhydramine
Drug: Placebo — Placebo matched to diphenhydramine 5% ointment
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate whether recruitment rates are adequate to power a future RCT. The secondary aims are to obtain preliminary information about safety and efficacy of topical diphenhydramine 5% ointment in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. ACR clinical criteria of knee OA
2. Radiographic knee OA (Kellgren-Lawrence grade >1)
3. Age ≥ 50 years
4. VAS pain >= 40/100 mm at baseline
5. Non-use of NSAIDs one week before the baseline
6. Symptoms present on most days for at least 3 months

Exclusion Criteria:

1. Any form of inflammatory arthritis
2. Use of another topical product at the application site
3. Treatment with intraarticular hyaluronic acid within 6 months
4. Treatment with intraarticular glucocorticoid within 2 months
5. Knee injury/surgery or diagnostic arthroscopy within 3 months
6. Allergic reaction to diphenhydramine or any component of the formulation
7. Participant has clinical signs and symptoms suggestive of COVID-19, eg, fever, dry cough, dyspnea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | through study completion, an average of 1 year
  Ability to recruit 8 patients per month

SECONDARY OUTCOMES:
Refusal rate | through study completion, an average of 1 year
  Number of eligible patients who refuse to participate
Adherence | through study completion, an average of 1 year
  Number of patients adhering to 80% of allocated treatment
Visual Analogue Scale for Pain | Baseline to week 1
  The Visual Analogue Scale for Pain varies from 0 to 10 cm. Higher values represent worse outcomes.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Pain | Baseline to week 1
  KOOS Pain consists of 9 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems..
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Symptoms | Baseline to week 1
  KOOS Symptoms consists of 7 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale Activities of daily living (ADL) | Baseline to week 1
  KOOS ADL consists of 17 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale of function in sports and recreation (Sport/Rec) | Baseline to week 1
  KOOS Sport/Rec consists of 5 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee injury and Osteoarthritis Outcome Score (KOOS) - subscale of quality of life (QOL) | Baseline to week 1
  KOOS QOL subscale of quality of life consists of 4 items, which are answered on a 4-point likert scale (0=no problems, 4=extreme problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Visual Analogue Scale for patient global assessment | Baseline to week 1
  The Visual Analogue Scale for patient global assessment varies from 0 to 10 cm. Higher values represent worse outcomes.
Global evaluation of treatment by patient | Baseline to week 1
  Global evaluation of treatment by patient on 5 point Likert scale. The Global Evaluation of treatment varies from 0 to 5. Higher values represent worse outcomes.
Percentage of patients achieving minimal clinically important improvement (MCII) of visual analogue scale (VAS) pain | Week 1
  Percentage of patients achieving MCII of VAS pain. The cut-off for MCII changes will be 15 of 100 for absolute improvement and 20% for relative improvement
Percentage of patients achieving minimal clinically important improvement (MCII) of visual analogue scale (VAS) patient's global assessment | Week 1
  Percentage of patients achieving MCII of VAS patient's global assessment The cut-offs for MCII changes will be 15 of 100 for absolute improvement and 20% for relative improvement for patient's global assessment
Percentage of patients achieving minimal clinically important improvement (MCII) of Knee injury and Osteoarthritis Outcome Score (KOOS) function of daily living | Week 1
  Percentage of patients achieving MCII of Knee injury and Osteoarthritis Outcome Score (KOOS) subscale of function of daily living.
  The cut-offs for MCII changes will be 8 of 100 for absolute improvement for KOOS function in daily living subscale score
Adverse events | Baseline to Week 1
  Any adverse event occurred during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Clinical Immunopharmacology, Novosibirsk, Russia